CLINICAL TRIAL: NCT06989021
Title: CORRELATION BETWEEN HAND, PINCH GRIP STRENGTH, WRIST JOINT POSITION SENSE AND FORWARD HEAD POSTURE AMONG DENTISTS
Brief Title: Forward Head Posture and Hand Function in Dentists
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hadeer E mohamed mohamed sharf el-deen, Hadeer Essam Mohamed, Cairo University
Other Study IDs: (NO: P.T.REC/012/005800)
Record Dates: First submitted 2025-05-17; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Forward Head Posture
Keywords: Craniovertebral Angle Hand Function Posture Assessment Wrist Proprioception

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational study investigates the correlation between forward head posture and hand grip strength, pinch grip strength, and wrist joint position sense among dentists aged 23-30 years. The aim is to understand the impact of poor head posture on upper limb function in dental professionals.

DETAILED DESCRIPTION:
The study evaluates the relationship between craniovertebral angle and upper limb strength and proprioception using hand dynamometers, pinch gauges, and goniometers. Forward head posture is assessed photometrically. A total of 82 participants will be recruited, all dentists, aged 23-30 years, with FHP confirmed by CVA <50°. Hand grip, pinch grip (tip, palmar, lateral), and wrist joint position sense (flexion/extension) will be assessed in the dominant hand only.

ELIGIBILITY:
Inclusion Criteria:

* Male and female dentists

Aged 23-30

BMI 18.5-29.9 kg/m²

Dominant hand used for testing

Forward head posture (CVA < 50°)

Exclusion Criteria:

* History of cervical trauma or surgery

Cervical radiculopathy or disc herniation

Upper limb neurological or orthopedic disorders

Dizziness, blurred vision, or neck/shoulder pain

Ages: 23 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Male and female dentists aged 23-30 years, including residents, interns, and senior dental students, with forward head posture (craniovertebral angle < 50°), recruited from the Faculty of Dentistry at Kafr El-Sheikh University. Participants must have a BMI between 18.5 and 29.9 kg/m² and no history of neurological or orthopedic disorders affecting the upper limb or cervical spine.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Hand Grip Strength | Single assessment at baseline
  To assess the strength of the dominant hand and examine its correlation with forward head posture (CVA < 50°).

SECONDARY OUTCOMES:
Pinch Grip Strength | Single assessment at baseline
  To assess the pinch grip strength of the dominant hand and evaluate its correlation with forward head posture.
Wrist Joint Position Sense | Single assessment at baseline
  To evaluate wrist joint proprioception and determine its association with forward head posture.

CONTACTS AND LOCATIONS:
Overall Officials: Hadeer Essam Mohamed, Bachelor's Degree, Principal Investigator — Cairo University; ENAS FAWZY YOUSSEF, PT, PhD, Study Chair — Cairo University

REFERENCES:
- [Background] Celik HI, Unver B, Akbas E, Erdem EU. Head posture mediates the association of cognition with hand grip and pinch strength in older adults: an examination using structural equation modeling. BMC Musculoskelet Disord. 2023 Apr 25;24(1):324. doi: 10.1186/s12891-023-06436-4. PMID 37098544